CLINICAL TRIAL: NCT06768931
Title: A Multicenter, Randomized Controlled Phase II Clinical Study of Standard Neoadjuvant Therapy Combined with Biolosion (oral Probiotic Compound Preparation) in Triple-negative Breast Cancer
Brief Title: Biolosion Combined Standard Neoadjuvant Therapy to Treat Triple-negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Mei-ting Chen, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-BC-PROBIOTIC
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer (TNBC); Early Stage Breast Cancer; Immunotherapy; Probiotic
Keywords: Triple negative breast cancer; Probiotics; Immunotherapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients in experimental group will be treated with standard neoadjuvant chemotherapy, immunotherapy combined with Biolosion (oral probiotic compound preparation). Patients in controlled group will be treated with standard neoadjuvant chemotherapy and immunotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Standard therapy (paclitaxel-carboplatin or docetaxel-carboplatin, and PD-1 antibody for 4 cycles followed by doxorubicin-cyclophosphamide or epirubicin-cyclophosphamide, and PD-1 antibody for 4 cycle) combined with compound preparation Biolosion
  Interventions: Other: Biolosion (oral probiotic compound preparation)
- Controlled group (No Intervention): Standard therapy, including paclitaxel-carboplatin or docetaxel-carboplatin, and PD-1 antibody for 4 cycles followed by doxorubicin-cyclophosphamide or epirubicin-cyclophosphamide, and PD-1 antibody for 4 cycle.

INTERVENTIONS:
Other: Biolosion (oral probiotic compound preparation) — Biolosion (oral probiotic compound preparation) will be administered in the experimental arm. Biolosion will be taken every night from day 1 to day 21 after each cycle of immunotherapy-chemotherapy.
  Arms: Experimental group

SUMMARY:
To evaluate the efficacy and safety of compound preparation Biolosion in combination with standard neoadjuvant therapy for locally advanced triple-negative breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 1.18 years and above, diagnosed with triple-negative breast cancer (ER≤10%, PR≤10%, HER-2 negative) by pathology;
2. Patients must have tumor specimens (formalin-fixed, paraffin-embedded, or fresh pre-treated tumor tissue) available for PD-L1 expression testing;
3. Researchers assess indications for neoadjuvant chemotherapy, with staging from IIA to IIIC, based on imaging or pathological evaluation of cT1c, N1-3, or cT2~cT4, cN0~N3, and patients with no distant metastasis as evaluated by imaging;
4. Patients must not have received chemotherapy or targeted therapy for advanced breast cancer;
5. ECOG PS: 0-2;
6. Expected survival of ≥12 weeks;
7. Major organ function levels must meet the following criteria:

1) Hematological examination standards must meet: ANC≥1.5×10^9/L, PLT≥75×10^9/L, Hb≥90g/L (no blood transfusions or blood products within 14 days, and no use of G-CSF or other hematopoietic growth factors for correction) 2) Biochemical examination must meet the following standards: TBIL<1.5×ULN, ALT, AST<2.5×ULN, for patients with liver metastasis, ALT, AST may be <5×ULN, BUN and Cr≤1×ULN or endogenous creatinine clearance ≥50ml/min (Cockcroft-Gault formula); 8. Women of childbearing age must have taken reliable contraceptive measures or undergone a pregnancy test (serum or urine) within 7 days prior to enrollment, with a negative result, and must be willing to use appropriate contraceptive methods during the trial and for 8 weeks after the last administration of the investigational drug.

9. Participants voluntarily join this study, demonstrate good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. There is a clear distant transfer;
2. A history of autoimmune diseases;
3. Acute or chronic active hepatitis B (defined as positive hepatitis B surface antigen and/or hepatitis B core antibody, with hepatitis B virus DNA copy number ≥1×10³ copies/ml or ≥200 IU/ml) or positive antibodies for acute or chronic active hepatitis C, with positive hepatitis C antibodies but negative RNA testing allowed for enrollment.
4. Previous treatment with immune checkpoint inhibitors;
5. Received systemic immunostimulants, systemic corticosteroids, or immunosuppressants within the last 4 weeks;
6. Any severe underlying disease, comorbidities, and active infections, or patients with severe metabolic disorders;
7. Currently receiving other antitumor treatments;
8. Known comorbidities (e.g., chronic diarrhea, inflammatory bowel disease, etc.) that, in the investigator's assessment, would increase the risk associated with the administration of the study drug or interfere with the interpretation of study results.
9. Currently using or planning to use probiotics, yogurt, or bacterial-enhanced foods during the treatment period.
10. A history of epilepsy or seizure-inducing states;
11. Pregnant or breastfeeding patients;
12. Poor compliance or inability to undergo normal follow-up;
13. Individuals allergic to the study drug;
14. Diagnosis of other malignancies within the past 5 years, with the exception of: surgically removed non-melanoma skin cancer, adequately treated cervical carcinoma in situ, locally curative prostate cancer, surgically treated ductal carcinoma in situ, or malignancies diagnosed 2 years prior to randomization without evidence of disease and untreated for ≤2 years;
15. The investigator's judgment on other conditions that may affect the conduct of the clinical study and the determination of study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2030-01-08 (Estimated); Study Completion 2035-02-08 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission | From enrollment to the end of treatment at 24 weeks
  ypT0N0, ypTisN0 after surgery

SECONDARY OUTCOMES:
overall survival | From enrollment to the end of treatment at 5 years
  The length of time from the date of the start of treatment until death.
Disease Free Survival | From enrollment to the end of treatment at 5 years
  Time from treatment until the recurrence of disease (or death) after undergoing curative-intent treatment.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Gansu Cancer Hospital, Lanzhou, Gansu
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Sun yat sen university cancer center, Guangzhou, Guangdong
  - Central Hospital of Guangdong Nongken, Zhanjiang, Guangdong
  - Zigong Fourth People's hospital, Zigong, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided